CLINICAL TRIAL: NCT01706341
Title: The Effect of Administering a Small Dose of Glucose on the Pregnant Women and Their Neonates During Cesarean Section
Brief Title: The Effect of Administering a Small Dose of Glucose During Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nagoya City University (Other)
Responsible Party: Principal Investigator, Yoshihito Fujita, MD, Associate professor, the department of Anesthesiology, Nagoya City University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCU-573
Record Dates: First submitted 2012-10-08; First posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Cesarean Section
Keywords: cesarean section; intravenous fluid; a glucose-containing solution; fetal hypoglycemia; neonatal hypoglycemia
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acetate Ringer's solution (Active Comparator): Administering acetate Ringer's solution that contains no glucose as an initial infusion A total infusion volume of acetate Ringer's solution is 1500ml
  Interventions: Drug: administer acetate Ringer's solution; Drug: acetate Ringer's solution containing no glucose
- acetate Ringer's solution with 1% glucose (Active Comparator): Administering the acetate Ringer's solution that contains 1% glucose as an initial infusion A total infusion volume of the acetate Ringer's solution containing 1% glucose is 1500ml (containing 15g of glucose)
  Interventions: Drug: administer acetate Ringer's solution; Drug: acetate Ringer's solution containing 1% glucose

INTERVENTIONS:
Drug: administer acetate Ringer's solution — During cesarean section under spinal anesthesia, each acetate Ringer's solution is administered before delivery.
Drug: acetate Ringer's solution containing no glucose
  Arms: acetate Ringer's solution
Drug: acetate Ringer's solution containing 1% glucose
  Arms: acetate Ringer's solution with 1% glucose

SUMMARY:
The purpose of this study is to investigate the effect of administering a small dose of glucose on the pregnant women and their neonates during cesarean section. We investigate the safety and efficacy of use of a glucose-containing solution for the pregnant women and the neonates.

DETAILED DESCRIPTION:
Rapid infusion of large amount of glucose is associated with fetal hyperglycemia, hyperinsulinemia, and neonatal hypoglycemia. However, the effect of small dose of glucose is unclear. We conducted a pilot study of small dose of glucose. We investigated the effect of a glucose-containing fluid on the blood sugar of the umbilical artery. We found that in the case of no-glucose-containing fluid, there were some cases in which umbilical arterial concentration of glucose was less than 50 mg/dl, which might cause neonatal hypoglycemia. In addition, in the case of 1%-glucose-containing fluid, mean umbilical arterial concentration of glucose was 97 mg/dl.

The purpose of this study is to investigate the effect of administering a small dose of glucose on the pregnant women and their neonates during cesarean section. We investigate the safety and efficacy of use of a glucose-containing solution for the pregnant women and the neonates.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cesarean section who met the criteria of the American Society of Anesthesiologists physical status of 1-2

Exclusion Criteria:

* ASA physical status >=3, Obesity (BMI>35), Height>=175cm, Weight>=80Kg

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
The blood glucose concentration in the neonates at one hour of age | One hour of age

SECONDARY OUTCOMES:
The blood glucose concentration in the neonates at two hour of age | Two hour of age

OTHER OUTCOMES:
Evidence of clinical complications (especially, low glucose symptoms) | Within the first 3 days after cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihito Fujita, MD. PhD., Study Chair — Department of Anesthesiology, Nagoya City Universtiy
Locations (1):
- Departiment of Anesthesiology, Nagoya City University Hospital, Nagoya, Japan